CLINICAL TRIAL: NCT05953467
Title: Healthcare Seeking Behavior of Frequent Emergency Care Visitors
Acronym: FEC
Status: Recruiting | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: METC Z20230010
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Emergency Care; Acute Care Chain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, observational. — None, observational study

SUMMARY:
This retrospective study is part of a research line from Zuyderland Medical Centre focusing on the acute care chain. The aim of the study is to focus on the frequent visitors of the Emergency Department (ED) and bridge the gap to out-of-hours primary care.

Although the Dutch healthcare system is unique with their 24/7 accessibility to primary care, crowding within the acute care chain is a growing problem, even in the Netherlands. Patients visiting an ED multiple times a year, the so called frequent visitors are one of the contributing factors of ED crowding. This relatively small group of patients accounts for a disproportionate number of many ED visits. In the United States, it is estimated that between 4.5 and 8% of patients are responsible for almost one third of the total annual number of ED visits, by visiting the ED four or more times per year. Dutch research by vd Linden found that 0.5% of total ED patients visited their ED frequently, however, they defined frequent visitors using a threshold of 7 visits per year. In our study, the cutoff of more than four visits per year to define a frequent visitor is used.

This study aims to gain insight in who Dutch frequent visitors are, or - in other words - what their baseline characteristics are, which complaints are responsible for their healthcare seeking behavior, and do these patients also seek medical help at other places during out-of-hours like a General Practitioner Cooperative (GPC)?

Existing ED and GCP data will be used to identify patients who either visited the ED or one of the adjacent GPCs 4 times or more in one year. Using these data, this study aims to answer the following questions:

Primary objective:

- How many patients present to the ED of the Zuyderland hospital in Heerlen and Sittard 4 times or more a year and what are the characteristics of these frequent visitors of the ED?

Secondary objective:

* How many patients present to the GPC of South East Limburg 4 or more times a year and what are their characteristics of frequent visitor?
* Is there an association between the characteristics of frequent visitors of the ED of the Zuyderland hospital and subsequent (frequent) presentation at the GPC?

DETAILED DESCRIPTION:
This study is a retrospective observational analysis of all patients aged 18 years or older at time of first presentation during the inclusion period, and who visited the ED of the Zuyderland or the GPC of Sittard-Geleen or Heerlen in the Netherlands between 1 January 2022 and 31 December 2022 and visited the ED or GPC 4 times or more during this year.

All patients presenting at the ED or GPC of Zuyderland Medical Center between 1 January 2022 and 31 December 2022, with an age of 18 years or older at time of first presentation during the inclusion period, will be included. Frequent visitors, defined as patients visiting the ED or GPC 4 times or more during these 12 months, will be identified and characterized.

The geography of south east Limburg and the locations of EDs with integrated GPC, ensure that visitors in general visit the same location.

All patients aged 18 years or older at first ED presentation in 2022 will be screened.

Data will be automatically extracted from a digital information system with a retrospective review of patients who visited the ED more than four times in 2022.

Informed consent procedure is not required in this study type (see Data Management).

Patients who have previously stated to the hospital that their data may not be used for scientific research will be excluded.

Data will be extracted from an existing database, providing a retrospective review of all ED and GPC patients. For this study, patients who visited our ED or GPC more than four times in the preceding 12 months will be included. Data will subsequently be collected from their hospital and GPC files and will be anonymized.

Descriptive statistics will be used to present the results. Differences in variables will be statistically analyzed using SPSS. Statistical tests will be chosen dependent on the number of included patients: Chi Square and Fisher Exact tests will be used with a significance p<0.05.

The following data/variables will be extracted from all patients:

* Age (at first ED or GPC visit during 2022)
* Sex
* Social security number (BSN), which only will be used to link the visitors of the ED and GPC
* Zip code area (only numbers)
* Medical history (chronical pain, oncological, heart/vascular disease, diabetes, psychiatric)
* Service characteristics (date, time of the day (day 8.00-17.00, evening 17.00-24.00), night (24.00-8.00))
* Presenting complaints

Data extracted specifically from ED patients:

* Number of ED visits during inclusion period.
* Triage category (according to the Manchester Triage System: 1-5)
* Mode of referral
* Mode of transportation to hospital (including dispatch center triage urgency)
* Destination: discharge, admission (including type of ward), referral to other clinic, death, leaving without seeing a physician.
* Presenting specialty
* Treating specialism

Data extracted specifically from GPC patients:

* Number of overall visits in 2022
* Urgency level at GPC
* Type of contact: visit, (telephone) consultation
* Treatment given at the GPC
* Referral to secondary care
* Time of contact (evening, night, weekend)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 years or older at first ED presentation in 2022 who visited the ED 4 times or more in 2022.
* All adult patients aged 18 years or older at first GPC presentation in 2022 who visited the GPC 4 times or more.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the ED or GPC of Zuyderland Medical Center between 1 January 2022 and 31 December 2022, with an age of 18 years or older at time of first presentation during the inclusion period, will be included. Frequent visitors, defined as patients visiting the ED or GPC 4 times or more during these 12 months, will be identified and characterized.
  The geography of south east Limburg and the locations of EDs with integrated GPC, ensure that visitors in general visit the same location.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
How many patients present to the ED of the Zuyderland hospital in Heerlen and Sittard 4 times or more a year and what are the characteristics of these frequent visitors of the ED? | 1 year
  Frequency count: Measure the exact number of ED visits for each patient over the specified time frame. Frequency count on the number of males and females. Frequency count on presenting complaints.

SECONDARY OUTCOMES:
How many patients present to the GPC of South East Limburg 4 times or more a year and what are their characteristics of frequent visitor? | 1 year
  Frequency count: Measure the exact number of GPC visits for each patient over the specified time frame. Frequency count on the number of males and females. Frequency count on presenting complaints.
Do frequent visitors of the ED visit the GPC frequently as well? | 1 year
  Calculate a correlation coefficient (e.g., Pearson's correlation) between the frequency of ED visits and GPC visits.
Do frequent visitors of the GPC visit the ED frequently as well? | 1 year
  Calculate a correlation coefficient (e.g., Pearson's correlation) between the frequency of ED visits and GPC visits.
Do frequent visitors of the ED and the GPC visit those for the same reason? | 1 year
  Compare the reasons of presenting at the ED with reasons on presenting to the GPC with a utilization ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No